CLINICAL TRIAL: NCT01221961
Title: A Study to Determine the Agreement Between Masimo Monitor and Standard of Care
Brief Title: Masimo Radical-7 Monitor a Useful Adjuvant During Major Spine Surgery
Status: Terminated | Type: Observational
Why Stopped: We completed the 62% of the cases, enough data to get a conclusion of the study.
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Principal Investigator, Ronald Wender, Chair of the anesthesia department, Cedars-Sinai Medical Center
Other Study IDs: Pro00021287
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Major Spine Surgery Procedure
Keywords: Major spine surgery; Hemoglobin; Blood transfusion

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Masimo Radical-7 — The Masimo device will be placed on one finger of the patient. To see whether or not the hemoglobin values recorded at the same time matches between the standard clinical practice (CSMC Lab and outside Lab) and the Masimo device

SUMMARY:
This is a study designed to compare the agreement of hemoglobin (Hb) measurements, documented at specific time points (the time a blood sample was obtained by the standard clinical care after physician/nurse orders it and, during that same time, the Hb value recorded by the Masimo Radical-7 monitor); recorded several times throughout patient's major spine surgery procedure (depending on how many times the physician/nurse orders the Hb value to be tested), between the standard clinical practice {intermittent measure of Hb [Cedar Sinai Medical Center (CSMC) Lab and outside lab) and Masimo radical-7 device (continuous, non-invasive Hb level measurements)*.

DETAILED DESCRIPTION:
*See whether or not the hemoglobin values recorded at the same time matches between the standard clinical practice (CSMC Lab and outside Lab) and the Masimo device

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo multiple level spine surgery procedures
* 18 - 80 years of age
* American Society of Anesthesiologists (ASA) Class I - III adults of either sex
* Pregnant women

Exclusion Criteria:

* Patients with a perfusion index less than 1 or low confidence reading
* Patients with nail polish and /or a nail deformity on a finger that would used for sensor placement
* Patient undergoing cardio-pulmonary bypass

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major spine surgery
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2010-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Hemoglobin value | 0-8 hours
  During the time surgery last.

SECONDARY OUTCOMES:
Blood transfusion | 0-8 hours
  During the time surgery last.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald H Wender, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical center, Los Angeles, California, United States